CLINICAL TRIAL: NCT05362084
Title: Comparison of Intravascular Injection Incidences Durig Lumbar Medial Branch Block Using Anteroposterior or Oblique Angle
Brief Title: Intravascular Injection Incidences During Lumbar Medial Branch Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-07-014-002
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Intravascular Injection
Keywords: intravascular injection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oblique group (Active Comparator): medial branch block with oblique group
  Interventions: Procedure: lumbar medial branch block
- Anteroposterior group (Placebo Comparator): medial branch block with anteroposterior group
  Interventions: Procedure: lumbar medial branch block

INTERVENTIONS:
Procedure: lumbar medial branch block — lumbar medial branch block

SUMMARY:
The purpose of this study is to compare using oblique fluoroscopic angle has any advantage in reducing the incidence of vascular punture and technical easiness during lumbar medial branch block

DETAILED DESCRIPTION:
In previous report, the use of oblique fluoroscopic angle during S1 transforaminal injection demonstrated technical easiness and reduced intravascular injection incidences. For the procedure lumbar medial branch block, both anteroposterior and oblique fluoroscopic angle are possible. Usually, which approach method to use is determined according to the physician's preferences.

The final target for lumbar medial branch block is the junction betweeen superior articular process and transverse process. This target can be easily confirmed under the scotty dog appearance. If we use oblique fluoroscopic angle, this approach (30 degree) can make scotty dog appearance more visible so that physician can identify bony landmark more easily for lumbar medial branch block. For beginners, oblique fluoroscopic approach seems to provide more advantages in identifying bony landmark. However, it is uncertain whether this approach can provide technicaL easiness and reduce the intravascualr injection incidences.

ELIGIBILITY:
Inclusion Criteria:

* facet joint arthropathy

Exclusion Criteria:

* allergy to local anesthetics or contrast medium
* pregnancy
* spine deformity
* neurologic abnormality

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
incidence of intravasuclar injection | 1 minute after finishing lumbar medial branch block
  incidence of intravasuclar injection

SECONDARY OUTCOMES:
time required to complete lumbar medial branch block | 1 second after finishing lumbar medial branch block
  time required to complete lumbar medial branch block
radiation amount to complete lumbar medial branch block | 1 second after finishing lumbar medial branch block
  radiation amount to complete lumbar medial branch block

CONTACTS AND LOCATIONS:
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No